CLINICAL TRIAL: NCT04369183
Title: Efficacy and Safety of Rituximab in Adult Patients With Refractory or Relapsed Primary Focal Segmental Glomerulosclerosis or Minimal Change Disease
Brief Title: Rituximab for Refractory or Relapsed Focal Segmental Glomerulosclerosis or Minimal Change Disease
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Mirioglu, Principal Investigator, Istanbul University
Other Study IDs: 2019/977
Record Dates: First submitted 2020-04-25; First posted 2020-04-30 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: Focal Segmental Glomerulosclerosis; Minimal Change Disease
Keywords: focal segmental glomerulosclerosis; minimal change disease; rituximab
MeSH Terms: conditions — Glomerulosclerosis, Focal Segmental; Nephrosis, Lipoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with primary focal segmental glomerulosclerosis or minimal change disease who were treated using rituximab (375 mg/m2/wk for 1-4 weeks) following resistance to or relapse after at least one set of prior therapies including corticosteroids, calcineurin inhibitors or mycophenolic acid derivatives.

SUMMARY:
Various studies have been conducted to identify effective treatment strategies for primary focal segmental glomerulosclerosis (FSGS) and minimal change disease (MCD) so far. In the light of these studies, corticosteroids and calcineurin inhibitors have been the treatment of choice and mycophenolic acid derivatives have been seen as a second line agent. However, treatment options in refractory or relapsed cases are still under debate. Recently, rituximab has become an alternative in those patients. Therefore, a study based on registry data was conducted to evaluate the efficacy and safety of rituximab in adult patients suffering from a relapsed or refractory primary FSGS or MCD.

ELIGIBILITY:
Inclusion Criteria:

* Having biopsy-proven focal segmental glomerulosclerosis or minimal change disease.
* Showing resistance to or relapsing after at least one set of prior therapies including corticosteroids, calcineurin inhibitors or mycophenolic acid derivatives.
* Having a history of rituximab use (375 mg/m2/wk for 1-4 weeks) following resistance to or relapse after aforementioned agents.

Exclusion Criteria:

* Not providing or withdrawing consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary focal segmental glomerulosclerosis or minimal change disease who were treated using rituximab following resistance to or relapse after at least one set of prior therapies including corticosteroids, calcineurin inhibitors or mycophenolic acid derivatives.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Complete Remission | 12 months
  Proteinuria <0.5 g/day, confirmed by two values at least 1 week apart, accompanied by a normal serum albumin concentration, and a normal serum creatinine.
Partial Remission | 12 months
  Proteinuria <3.5 g/day and a 50% or greater reduction from peak values, confirmed by two values at least 1 week apart, accompanied by an improvement or normalization of the serum albumin concentration and stable serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Yazici, MD, Study Chair — Department of Internal Medicine, Istanbul Faculty of Medicine; Safak Mirioglu, MD, Principal Investigator — Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruggenenti P, Ruggiero B, Cravedi P, Vivarelli M, Massella L, Marasa M, Chianca A, Rubis N, Ene-Iordache B, Rudnicki M, Pollastro RM, Capasso G, Pisani A, Pennesi M, Emma F, Remuzzi G; Rituximab in Nephrotic Syndrome of Steroid-Dependent or Frequently Relapsing Minimal Change Disease Or Focal Segmental Glomerulosclerosis (NEMO) Study Group. Rituximab in steroid-dependent or frequently relapsing idiopathic nephrotic syndrome. J Am Soc Nephrol. 2014 Apr;25(4):850-63. doi: 10.1681/ASN.2013030251. Epub 2014 Jan 30. PMID 24480824